CLINICAL TRIAL: NCT05223972
Title: The Comparasion Effect of Lyon and Schroth Techniques on Adolescent İdiopathic Scoliosis
Brief Title: Effect of Lyon and Schroth Techniques on Adolescent İdiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Mehmet Hanifi Kaya, lecturer, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27.04.2021-10774
Record Dates: First submitted 2022-01-12; First posted 2022-02-04 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scoliosis Treatment Group (Experimental): For the scoliosis group treatment include schroth theraphy
  Interventions: Other: Schroth Treatment
- Lyon Treatment (Experimental): For the scoliosis group treatment include Lyon theraphy..
  Interventions: Other: Schroth Treatment

INTERVENTIONS:
Other: Schroth Treatment — Schroth exercises consist of passive and active postural auto-correction exercises done repeatedly and based on kinesthetic and sensorimotor principles. The ultimate goal of the Schroth method is to enable the patient to consciously maintain correct posture in their daily living activities. To achieve this requires repeating corrective movements performed to improve postural motor control. Schroth exercises also include strength and endurance training of postural muscles in order to improve the curve, raise the patient's self-image, and reduce pain. In this study, the Schroth exercises progressed from more to less passive support, from more to less feedback, and from lying to sitting or standing positions, according to the patient's ability to perform the specific exercise
  Other Names: Lyon Treatment

SUMMARY:
Today, it is known that the conservative treatment of scoliosis is gaining importance. In addition, no study has been found comparing the efficacy of two important conservative treatment methods, the Schroth and Lyon method, in adolescent idiopathic scoliosis. Accordingly, this study was conducted to compare the effectiveness of schroth and Lyon exercises in individuals with AIS.

ELIGIBILITY:
Inclusion Criteria:

* Participants were between ages 10-18,
* Volunteered for the study,
* Diagnosed with adolescent idiopathic scoliosis,
* Cobb angle between 10-30 degrees,
* 0-3 Risser sign,
* Sanders classification 0-4 ,
* Lenke curve type 1

Exclusion Criteria:

* Participants who other type of scoliosis
* Previous spinal surgery
* Exercise contraindications
* Rheumatological disease
* Another neuromuscular problem were excluded from the study.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-06-12 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Cobb angle | 6 months
  Cobb measurement

SECONDARY OUTCOMES:
Scoliosis research society-22 | 6 months
  Quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Turkey (Türkiye)